CLINICAL TRIAL: NCT02199392
Title: A Pharmacokinetic Study to Assess the Influence of P-glycoprotein Inhibition and Simultaneous CYP3A4 and P-glycoprotein Induction on E7080 Pharmacokinetics Following Single Dose Oral Administration of 24 mg E7080 to Healthy Volunteers
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Eisai Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: E7080-A001-007
Record Dates: First submitted 2014-07-22; First posted 2014-07-24 (Estimated); Last update posted 2015-02-16 (Estimated); Status verified 2015-01

CONDITIONS: P-glycoprotein; Healthy Volunteers
Keywords: P-glycoprotein; Healthy Volunteers
MeSH Terms: interventions — lenvatinib

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Lenvatinib 24 mg (Experimental): The Pretreatment Phase will have two periods: Screening and Baseline 1. The Treatment Phase will have three periods: Treatment Period 1, Treatment Period 2, and Treatment Period 3 with a Baseline 2 assessment prior to Treatment Period 2 and a Baseline 3 assessment prior to Treatment Period 3. In the Treatment Phase, subjects will take a single oral dose of 24 mg lenvatinib on three separate occasions (Period 1, Day 1; Period 2, Day 15; and Period 3, Day 43). In Period 2, Day 15, subjects will also take a single oral dose of 600 mg po rifampin. In Period 3, subjects will receive 600 mg rifampin po daily for 21 days (Period 3, Days 29 to 49). On Day 43 of Period 3, subjects will take 24 mg lenvatinib in addition to the rifampin.
  Interventions: Drug: Lenvatinib

INTERVENTIONS:
Drug: Lenvatinib — subjects will take a single oral dose of 24 mg lenvatinib on three separate occasions (Period 1, Day 1; Period 2, Day 15; and Period 3, Day 43). In Period 2, Day 15, subjects will also take a single oral dose of 600 mg po rifampin. In Period 3, subjects will receive 600 mg rifampin po daily for 21 days (Period 3, Days 29 to 49). On Day 43 of Period 3, subjects will take 24 mg lenvatinib in addition to the rifampin.
  Other Names: E7080

SUMMARY:
The purpose of this single-dose, open-label, sequential, three-period study in 15 healthy subjects was to assess the influence of P-glycoprotein inhibition and simultaneous CYP3A4 and P-glycoprotein induction on lenvatinib pharmacokinetics following single dose oral administration of 24 mg lenvatinib to healthy volunteers.

DETAILED DESCRIPTION:
This is a single-dose, open-label, sequential, three-period study in 15 healthy subjects to assess the influence of P-glycoprotein inhibition and simultaneous CYP3A4 and P-glycoprotein induction on lenvantinib pharmacokinetics following single dose oral administration of 24 mg lenvatinib to healthy volunteers. The study will consist of two phases: Pretreatment and Treatment. The Pretreatment Phase will have two periods: Screening and Baseline 1. The purpose of the Screening Period is to obtain informed consent and to establish protocol eligibility. The purpose of the Baseline 1 is to confirm protocol eligibility. The Treatment Phase will have three periods: Treatment Period 1, Treatment Period 2, and Treatment Period 3 with a Baseline 2 assessment prior to Treatment Period 2 and a Baseline 3 assessment prior to Treatment Period 3. The purpose of Baselines 2 and 3 are to confirm continued protocol eligibility. In the Treatment Phase, subjects will take a single oral dose of 24 mg lenvatinib on three separate occasions (Period 1, Day 1; Period 2, Day 15; and Period 3, Day 43). In Period 2, Day 15, subjects will also take a single oral dose of 600 mg po rifampin. In Period 3, subjects will receive 600 mg rifampin po daily for 21 days (Period 3, Days 29 to 49). On Day 43 of Period 3, subjects will take 24 mg lenvatinib in addition to the rifampin.

ELIGIBILITY:
Inclusion Criteria

Subjects must meet all of the following criteria to be included in this study:

1. Non-smoking (i.e., no use of nicotine or nicotine containing products within the past 3 months), male or female subjects, age greater than or equal to 18 years and lesser than or equal to 55 years
2. Body mass index (BMI) greater than or equal to 18 and lesser than or equal to 30 kg/m2 at Screening
3. Females may not be lactating or pregnant at Screening or Baseline (as documented by a negative beta-human chorionic gonadotropin [B-hCG] test with a minimum sensitivity of 25 IU/L or equivalent units of B-hCG). A separate baseline assessment is required if a negative screening pregnancy test was obtained more than 72 hours before the first dose of study drug
4. All females will be considered to be of childbearing potential unless they are postmenopausal (amenorrheic for at least 12 consecutive months, in the appropriate age group, and without other known or suspected cause) or have been sterilized surgically (i.e., bilateral tubal ligation, total hysterectomy, or bilateral oophorectomy, all with surgery at least 1 month before dosing)
5. Females of childbearing potential must not have had unprotected sexual intercourse within 30 days prior to study entry and must agree to use a highly effective method of contraception (e.g., total abstinence, a nonhormonal-based intrauterine device, a doublebarrier method [such as condom plus diaphragm with spermicide], or have a vasectomised partner with confirmed azoospermia) throughout the entire study period and for 30 days after study drug discontinuation. Use of hormonal contraceptives (e.g., oral contraceptive, contraceptive implant, hormone-releasing IUD) as the primary method of contraception does not meet the definition of a highly effective method of birth control for this study because Rifampin is known to cause failure of hormonal contraceptives. If currently abstinent, the subject must agree to use a double-barrier method as described above if she becomes sexually active during the study period or for 30 days after study drug discontinuation
6. Male subjects must have had a successful vasectomy (confirmed azoospermia) or they and their female partner must meet the criteria above (i.e., not of childbearing potential or practicing highly effective contraception throughout the study period and for 30 days after study drug discontinuation). No sperm donation is allowed through the study period and for 30 days after study drug discontinuation
7. Provide written informed consent
8. Are willing and able to comply with all aspects of the protocol

Exclusion Criteria

Subjects who meet any of the following criteria will be excluded from this study:

1. Subjects who had a clinically significant illness that required medical treatment within 8 weeks or a clinically significant infection within 4 weeks of dosing
2. Subjects with a disease that may influence the outcome of the study; such as psychiatric disorders and disorders of the gastrointestinal tract, liver, kidney, respiratory system, endocrine system, hematological system, neurological system, or cardiovascular system, or subjects who have a congenital abnormality in metabolism within 4 weeks prior to dosing
3. Subjects with a history of gastrointestinal surgery (hepatectomy, nephrotomy, digestive organ resection, etc.) that may affect pharmacokinetic profiles of lenvatinib or rifampin
4. Subjects with a known history of clinically significant drug or food allergies or presently experiencing significant seasonal allergy
5. Subjects who experienced a weight loss or gain of more than 10% between Screening and prior to dosing
6. Subjects with any clinically abnormal symptom or organ impairment found on medical history, symptoms/signs, vital signs, ECG finding, or laboratory test results which require medical treatment
7. Subjects with a QTc interval greater than 450 ms at Screening or Baseline
8. Subjects with a hemoglobin level lesser than 12.0 g/dL
9. Subjects who had a positive result from human immunodeficiency virus (HIV) or hepatitis C virus antibody (HCVAb) screening tests, or clinical evidence of active viral hepatitis A or B
10. Subjects with a known or suspected history of drug or alcohol misuse within 6 months prior to Screening, or a positive urine drug or alcohol test at Screening or Baseline
11. Subjects who have consumed caffeinated beverages within 72 hours prior to Baseline
12. Subjects who have taken dietary supplements, juice, or herbal preparations or other foods or beverages that may affect various drug metabolizing enzymes and transporters [e.g., alcohol, grapefruit, grapefruit juice, grapefruit-containing beverages, apple or orange juice, vegetables from the mustard green family (e.g., kale, broccoli, watercress, collard greens, kohlrabi, brussel sprouts, mustard), and charbroiled meats] within 2 weeks prior to dosing
13. Subjects who have taken herbal preparations containing St. John's Wort within 4 weeks prior to dosing
14. Subjects who have taken prescription drugs within 4 weeks prior to dosing
15. Subjects who have taken over-the-counter (OTC) medications within 2 weeks prior to dosing
16. Subjects who have participated in another clinical trial of an investigational drug or device within 4 weeks prior to dosing
17. Subjects who have received blood products within 4 weeks, or donated blood within 8 weeks, or donated plasma within 1 week of dosing
18. Subjects who have engaged in heavy exercise within 2 weeks prior to dosing (e.g., marathon runners, weight lifters, etc.)
19. Subjects who have any condition that would make him/her, in the opinion of the investigator, unsuitable for the study or who, in the opinion of the investigator, are not likely to complete the study for any reason
20. Known intolerance to the study drugs or any of the excipients
21. Females who are either pregnant or lactating

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 15 (Actual)
Dates: Start 2011-11; Primary Completion 2012-01 (Actual); Study Completion 2012-01 (Actual)

PRIMARY OUTCOMES:
Pharmacokinetics of lenvatinib: Cmax | Predose and up to 168 hours post dose
Pharmacokinetics of lenvatinib: AUC(0-inf) | Predose and up to 168 hours post dose

SECONDARY OUTCOMES:
Pharmacokinetics of lenvatinib: AUC(0-inf) | Predose and up to 168 hours post dose
Safety as measured by all Adverse Events (AEs) | Predose and up to 168 hours post dose
Safety as measured by laboratory values | Predose and up to 168 hours post dose
Safety as measured by physical examinations | Predose and up to 168 hours post dose
Safety as measured by vital signs | Predose and up to 168 hours post dose
Safety as measured by ECGs | Predose and up to 168 hours post dose

CONTACTS AND LOCATIONS:
Locations (1):
- Tacoma, Washington, United States